CLINICAL TRIAL: NCT02592408
Title: A Study to Assess Current Standard Malaria Treatment Guidelines and Evaluate Recently Developed G6PD Diagnostic Tools in the Republic of the Sudan
Brief Title: A Study to Assess Current Standard Malaria Treatment Guidelines in the Republic of the Sudan
Acronym: MalTreSu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: University of Khartoum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MenziesSHR
Record Dates: First submitted 2015-10-26; First posted 2015-10-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pf: ASP (Active Comparator): In falciparum patients (Pf): 3 days of artesunate + sulfadoxine/pyrimethamine (ASP)
  Interventions: Drug: ASP
- Pv: ASP + 14DPQ on day 2 (Active Comparator): In vivax patients (Pv): 3 days of artesunate + sulfadoxine/pyrimethamine (ASP) and 14 days of primaquine (14DPQ) starting on day 2
  Interventions: Drug: ASP; Drug: 14DPQ
- Pf: ASP + SDPQ (Active Comparator): In falciparum patients (Pf): 3 days of artesunate + sulfadoxine/pyrimethamine (ASP) and a single dose of primaquine (SDPQ) on day 2
  Interventions: Drug: ASP; Drug: SDPQ
- Pv: ASP + 14DPQ on day 42 (Active Comparator): In vivax patients (Pv): 3 days of artesunate + sulfadoxine/pyrimethamine (ASP) and 14 days of primaquine (14DPQ) starting on day 42
  Interventions: Drug: ASP; Drug: 14DPQ on Day 42

INTERVENTIONS:
Drug: ASP — 3 days of artesunate sulfadoxine/pyrimethamine on days 0-2
Drug: SDPQ — single dose primaquine on day 2
  Arms: Pf: ASP + SDPQ
Drug: 14DPQ — 14 day primaquine starting on day 2
  Arms: Pv: ASP + 14DPQ on day 2
Drug: 14DPQ on Day 42 — 14 day primaquine starting on day 42
  Arms: Pv: ASP + 14DPQ on day 42

SUMMARY:
This is a randomized controlled trial to assess the efficacy and safety of the national malaria treatment guidelines, asses the efficacy and safety of artesunate and sulphadoxine - pyrimethamine (AS+SP) for treatment in uncomplicated P. falciparum and P. vivax malaria and the hematologic effect of 14 days routine primaquine based radical cure in patients suffering from a P. vivax or mixed infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 months
* P. vivax or P. falciparum mono-infection or P. vivax / P. falciparum mixed infection
* Presence of axillary temperature ≥ 37.5°C or history of fever during the past 24 hrs
* Able to tolerate oral medication
* Able and willing to comply with the study protocol for the duration of the study
* Informed consent from the patient or from a parent or guardian in the case of children

Exclusion Criteria:

* Bodyweight ≤5kg
* Presence of general danger signs in children aged under 5 years or signs of severe malaria in any patient according to the definitions of WHO
* Presence of severe malnutrition
* Acute anaemia <8g/dL
* Regular medication, which may interfere with antimalarial pharmacokinetics
* History of hypersensitivity reactions or contraindications to any of the drug(s) tested or used as alternative treatment(s)
* A positive pregnancy test or lactating.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The recurrence of parasitaemia within 42 days of follow in P. falciparum infections | In the first 42 days
  Outcome measure is presented unadjusted and adjusted for PCR and compared between P. falciparum intervention and control arm
The recurrence of parasitaemia within 42 days of follow in P. vivax infections | In the first 42 days
  Outcome measure is presented unadjusted and adjusted for PCR and compared between P. vivax intervention and control arm

SECONDARY OUTCOMES:
The proportion of patients with any parasitemia on day 1, 2 and 3 after treatment | on days 1,2,3
  Outcome measure is stratified for P. falciparum and P. vivax infections
The proportion of patients with fever on day 1, 2 and 3 after treatment | on days 1, 2, 3
  Outcome measure is stratified for P. falciparum and P. vivax infections
The proportion of patients with gametocytemia on any of the follow up dates | In the first 42 days
  Outcome measure is stratified for P. falciparum and P. vivax infections
The proportion of patients with severe anaemia (Hb<7g/dl) or requiring blood transfusion within 42 days of enrolment | In the first 42 days
  Outcome measure is stratified for P. falciparum and P. vivax infections
The fractional change in Hb between baseline and day 7,14 and 16 (incl. proportion of patients with >25% drop in Hb between the time points) in vivax / mixed infection patients receiving PQ | on days 0, 7, 14 and 16
  Outcome measure is stratified for P. falciparum and P. vivax infections
The proportion of patients with adverse and serious adverse events | In the first 42 days
  Outcome measure is stratified for P. falciparum and P. vivax infections
The proportion of vivax patients adhering to 14 days of primaquine treatment in the vivax cohort as measured by pill count | at the end of 14DPQ treatment (day 16)
The distribution of G6PD activity among the study population | on day of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Muzamil Mahdi, PhD, Principal Investigator — University of Khartoum
Locations (2):
- Sudan (2):
  - New Halfa Hospital, New Halfa, Kassalla
  - Gizeria Slang Hospital, Khartoum, Khartoum State

REFERENCES:
- [Derived] Hamid MMA, Thriemer K, Elobied ME, Mahgoub NS, Boshara SA, Elsafi HMH, Gumaa SA, Hamid T, Abdelbagi H, Basheir HM, Marfurt J, Chen I, Gosling R, Price RN, Ley B. Low risk of recurrence following artesunate-Sulphadoxine-pyrimethamine plus primaquine for uncomplicated Plasmodium falciparum and Plasmodium vivax infections in the Republic of the Sudan. Malar J. 2018 Mar 16;17(1):117. doi: 10.1186/s12936-018-2266-9. PMID 29548285